CLINICAL TRIAL: NCT05221450
Title: Factors Affecting the Endodontic Treatment Outcome
Status: Recruiting | Type: Observational
Sponsor: Odontos, Specialisticna Zobna Ambulanta, d.o.o. (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 0120-402/2019/5
Record Dates: First submitted 2022-01-22; First posted 2022-02-03 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Apical Periodontitis; Apical Granuloma; Apical Cyst
Keywords: root canal treatment; outcome; success
MeSH Terms: conditions — Periapical Periodontitis; Periapical Granuloma; Radicular Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: primary endodontic treatment
  Other Names: secondary endodontic treatment

SUMMARY:
The aim of this prospective cohort observational study is: (i) to assess the endodontic treatment outcome in a private specialist endodontic office in Slovenia; (ii) to estimate the effect of various pre-, intra- and postoperative factors onto endodontic treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to the private endodontic specialist office for endodontic treatment
* written informed consent was obtained prior beginning of the treatment.

Exclusion Criteria:

* preoperative advanced periodontal disease
* prior microsurgical root-end resection performed
* apices of the tooth were not clearly discernible on any of periapical radiographs
* endodontic treated teeth were extracted for non-endodontic reason
* the patient did not attend a follow-up examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample population will include patients who are referred from a general dental practices in Slovenia to a private specialist endodontic practice for endodontic treatment, from the beginning of January 2008 on. All patients will be over 18 years of age at the beginning of the endodontic treatment and will attent a follow-up examination at least 1-4 years after endodontic treatment.
  Teeth will not be included in the study if (i) they have preoperative advanced periodontal disease, (ii) prior microsurgical root-end resection was performed, or (iii) the apex / apices of the tooth are not clearly discernible on any of the periapical radiographs.
  Teeth will be excluded from the study if (i) they will be extracted for non-endodontic reason or (ii) the patient will not attend a follow-up examination.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome based on strict combined radiographic and clinical criteria | 1-4 years postoperatively
  Successful treatment outcome is defined as an absence of radiographic sign of apical periodontitis (periapical index PAI <= 2) and clinical signs of inflamation (swelling, sinus tract, tenderness to periapical palpation and percussion, pain) on follow-up examination 1-4 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Odontos, specialistična zobna ambulanta, d.o.o., Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
anonymised IPD that uderlie the results in the publication will we shared to other researcher on reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: anonymised data will be available on request for 1 year after the publication of the study report
Access Criteria: contacting the principal investigator by e-mail

REFERENCES:
- [Background] Ng YL, Mann V, Gulabivala K. A prospective study of the factors affecting outcomes of nonsurgical root canal treatment: part 1: periapical health. Int Endod J. 2011 Jul;44(7):583-609. doi: 10.1111/j.1365-2591.2011.01872.x. Epub 2011 Mar 2. PMID 21366626
- [Background] Friedman S, Abitbol S, Lawrence HP. Treatment outcome in endodontics: the Toronto Study. Phase 1: initial treatment. J Endod. 2003 Dec;29(12):787-93. doi: 10.1097/00004770-200312000-00001. PMID 14686806
- [Background] European Society of Endodontology. Quality guidelines for endodontic treatment: consensus report of the European Society of Endodontology. Int Endod J. 2006 Dec;39(12):921-30. doi: 10.1111/j.1365-2591.2006.01180.x. PMID 17180780
- [Background] Ng YL, Mann V, Rahbaran S, Lewsey J, Gulabivala K. Outcome of primary root canal treatment: systematic review of the literature - part 1. Effects of study characteristics on probability of success. Int Endod J. 2007 Dec;40(12):921-39. doi: 10.1111/j.1365-2591.2007.01322.x. Epub 2007 Oct 10. PMID 17931389
- [Background] Ng YL, Mann V, Rahbaran S, Lewsey J, Gulabivala K. Outcome of primary root canal treatment: systematic review of the literature -- Part 2. Influence of clinical factors. Int Endod J. 2008 Jan;41(1):6-31. doi: 10.1111/j.1365-2591.2007.01323.x. Epub 2007 Oct 10. PMID 17931388
- [Background] Ricucci D, Russo J, Rutberg M, Burleson JA, Spangberg LS. A prospective cohort study of endodontic treatments of 1,369 root canals: results after 5 years. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Dec;112(6):825-42. doi: 10.1016/j.tripleo.2011.08.003. PMID 22099859